CLINICAL TRIAL: NCT06720896
Title: Vision and Inflammation Study Testing Anti-acarid Therapeutics (VISTA-1): A Phase 2, Controlled, Double Blind, Randomized and Multicenter Study to Compare Efficacy and Safety of a Novel Topical Therapy (APT-001, Spinosad 1.8%) in Patients With Blepharitis.
Brief Title: A Phase 2, Controlled, Double Blind, Randomized and Multicenter Study to Compare Efficacy and Safety of a Novel Topical Therapy (APT-001, Spinosad 1.8%) in Patients With Blepharitis.
Acronym: VISTA-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aperta Biosciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VISTA-1
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Blepharitis
Keywords: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — spinosad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Active Comparator): APT-001 topical ophthalmic ointment, administered once daily for approximately 43 days
  Interventions: Drug: APT-001 topical ophthalmic ointment (spinosad)
- Control (Placebo Comparator): Vehicle control of APT-001 topical ophthalmic ointment, administered once daily for approximately 43 days
  Interventions: Drug: Vehicle control for APT-001 topical ophthalmic ointment

INTERVENTIONS:
Drug: APT-001 topical ophthalmic ointment (spinosad) — APT-001 topical ophthalmic ointment, administered once daily
  Arms: Active
Drug: Vehicle control for APT-001 topical ophthalmic ointment — Vehicle control for APT-001 topical ophthalmic ointment, administered once daily
  Arms: Control

SUMMARY:
The purpose of this study is to establish the clinical efficacy of APT-001 topical therapy 1.8% in patients with blepharitis as compared to its vehicle control, and to establish that the therapeutic is safe and generally well tolerated by patients.

DETAILED DESCRIPTION:
This Phase 2 study is a randomized, controlled, double-blind trial to compare the safety and efficacy of APT-001 1.8% to vehicle control for the treatment of blepharitis. The primary objective of the study is to compare the safety and efficacy of APT-001 compared to its vehicle from Day 1 to Day 43 in patients with blepharitis. The primary efficacy endpoint will be cure based upon collarettes. Safety will be determined by assessing adverse effects related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic blepharitis.
* At least 6 years of age.
* Eyelid collarette count (minimum score 2).
* Willing and able to follow all instructions and attend all study visits.
* Able to avoid prohibited medication for the duration of the study.
* Patients can willingly provide consent or have a legal authorized representative provide consent on the informed consent (IC) Form.

Exclusion Criteria:

* Women with confirmed pregnancies.
* Utilizing any current medical therapy for the eye.
* History of allergic reaction to spinosad or any formulation component.
* Patients using eyelid hygiene or other treatment(s) for blepharitis within 14 days of screening.
* History of ocular surgery within the past 1 year.
* Presence of other ocular diseases that may affect study outcomes (Corneal Dystrophies, Salzmanns disease, Severe dry eye, Keratoconus, Glaucoma filtering blebs).
* Use of investigational drug, chronic glaucoma medications, steroid.
* Uncontrolled systemic disease.
* Acute or chronic illness that would confound study results.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Collarette Cure | From enrollment to the end of treatment at 6 weeks
  Eyelid collarette count score 0

SECONDARY OUTCOMES:
Overall reduction in combined eyelid collarette and erythema scores | From enrollment to the end of treatment at 6 weeks
  Overall reduction in combined eyelid collarette and erythema scores
Erythema Cure rate | From enrollment to the end of treatment at 6 weeks
  Erythema Cure rate
Combined Cure rate | From enrollment to the end of treatment at 6 weeks
  Combined Cure rate
Demodex mite density | From enrollment to the end of treatment at 6 weeks
  Demodex mite density
Time to a Combined Cure. | From enrollment to the end of treatment at 6 weeks
  Time to a Combined Cure

CONTACTS AND LOCATIONS:
Overall Officials: Josue Moran, Ph.D., Study Director — Aperta Biosciences, LLC
Locations (2):
- Guatemala (2):
  - Dr. Rudy Gutierrez Diaz Sede Central, Guatemala City
  - EyeScan, Imágenes Diagnósticas Oculares, S. A., Guatemala City

IPD SHARING:
Plan to Share IPD: No